CLINICAL TRIAL: NCT01498432
Title: Phase 4, Single Centre, Single Blinded,Prospective Randomised Cross Over Comparison on the Physiological Response of Post Extubation Intensive Care Patients to Non-invasive Ventilation Using Either Air O2 or Heliox21
Brief Title: Physiological Response to Heliox21 and Air O2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 08/0339; 2009-009599-11 (EudraCT Number)
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heliox21 (Experimental)
  Interventions: Drug: Heliox21
- Air O2 (Active Comparator)
  Interventions: Drug: Air O2

INTERVENTIONS:
Drug: Heliox21 — For Heliox21 the percentage of O2 will match the percentage of O2 prior to extubation, and Helium will make up the remainder (e.g. Helium 65% + O2 35%), and the O2 concentration will be titrated as their clinical condition indicates (as O2 increases Helium will decrease and vice versa).
  Arms: Heliox21
Drug: Air O2 — For Air-O2 the percentage of O2 delivered will match the patient's percentage of O2 prior to extubation, and will be titrated as their clinical condition indicates.
  Arms: Air O2

SUMMARY:
This is a non-commercial study to explore the use of Heliox21 in a new patient cohort. The fundamental aim is to assess the therapeutic benefits of Heliox21 and practicalities of gas delivery in patients who require non-invasive ventilatory support following extubation on the Intensive Care Unit. Thus, the investigators aim to extend our knowledge of the potential role for Heliox21 in the post-extubation environment of the Intensive Care Unit. The purpose of this study is to answer a specific, clinically relevant question. That is whether Heliox21 helps to reduce the effort of breathing in the period following withdrawal of mechanically assisted ventilation in patients on the intensive care unit.

DETAILED DESCRIPTION:
Failure to wean from mechanical ventilatory support occurs when the magnitude of respiratory system loading exceeds its capacity to respond. Extubation success depends on the condition being resolved or improved. Gas exchange capacity, respiratory muscle strength, laryngeal function and cough strength, nutritional status and psychological state can all lead to extubation failure. However, efforts to reduce the work of breathing might offer an alternative strategy.

Studies recently carried out in both paediatric and adult populations disclose the serious consequences of failed extubation, namely prolonged intensive care and hospital stays, greater mortality rates and increased care costs.

Gas flow in an airway can be either laminar or turbulent. There needs to be a greater pressure differential to drive a turbulent flow than a laminar one. Helium is an inert gas with no systemic biological effects (at standard temperature and pressure).

The low density and viscosity of Helium means that its substitution for nitrogen in air allows laminar flow to be maintained at much higher flow rates, and flow rates to be maintained at much lower working pressures (5). As a result, the use of helium-oxygen mixtures (Heliox21) has potential to reduce work of breathing, and also to limit dynamic gas trapping through increased cavity emptying, and altered lung mechanics/ forced expiratory pressures. As a result, Heliox21 has been used as a respiratory therapeutic bridge for over 30 years, with demonstrable advantage in the management of conditions including tracheal obstruction and chronic obstructive pulmonary disease (COPD).

In theory, the use of Heliox21 should reduce work of breathing by improving the balance between work demand and capacity during the process of weaning patients from mechanical ventilation. In general studies of the use of Heliox21 after extubation have been limited. Thus, we aim to extend our knowledge of the potential role for Heliox21 in the post-extubation environment of the Intensive Care Unit. Whilst Heliox21 has generally been administered through a simple face-mask (+/- rebreathing bag), the development of the HAMILTON G5 AVEA ventilator now allows the accurate administration of Heliox21 (21% helium/79% oxygen) with defined inspired fractional oxygen concentrations. This advent offers the means to safely administer helium as an adjunct to non-invasive ventilatory support.

Main inclusion criteria:

All patients with a predicted requirement for post extubation non-invasive ventilatory support continuous positive airway pressure/bilevel positive airway pressure/noninvasive ventilation(CPAP/BiPAP/NIV) will be eligible.

The primary outcome measure:

The difference between the frequency to tidal volume (f/VT) ratio* after four hours of Heliox21 and the f/VT ratio after four hours of Air O2.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years
2. Males
3. Females
4. Any patient requiring mechanical ventilation for 5 days or more and/or has a tracheostomy to assist weaning from mechanical ventilation who has one or more of following risk factors suggesting that they are at risk of needing post extubation continuous positive airway pressure (CPAP), BiLevel positive airway pressure (BiPAP) or non-invasive ventilation (NIV):

   * BMI of 28 or more
   * Underlying respiratory disease (including asthma, COPD and bronchiectasis) as documented in medical notes for this current hospital admission.
   * SpO2 < 95% on 35% FiO2 or more
   * Smoker
   * Ex-smoker less than 12 months
   * Ex-smoker 10 pack year* or more history * Pack year = (Number of cigarettes per day X Number of years) ÷ 20

Exclusion Criteria:

1. Age < 18 years
2. Patient/legal representative refusal or inability to consent
3. Adults with learning disabilities/ dementia
4. Any contraindication to non-invasive ventilation:

   Inability to use mask (trauma/surgery) Excessive secretions Haemodynamic instability/life threatening arrhythmia
5. High risk of aspiration:

   * Impaired mental status (Detained under the Mental Health Act)
   * Un-co-operative/agitated patient
   * Life threatening refractory hypoxemia
   * Undrained pneumothorax
   * Bullae on X-Ray
   * Recent upper GI anastamosis
6. Patients already enrolled in an interventional
7. Females known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The difference between the f/VT ratio* | After four hours of Heliox21 and after four hours of Air O2.
  *f/VT is the measurement of breathing rate to tidal volume (f/VT) ratio

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hargreaves, Study Director — Whittington Hospital NHS Trust; Daniel S Martin, Principal Investigator — University College, London
Locations (1):
- Whittington Hospital NHS Trust, London, United Kingdom